CLINICAL TRIAL: NCT00221169
Title: Can PET CT Coregistration Imaging Adequately Determine the Gross Tumor Volume and Microscopic Extension in Non-Small Cell Lung Cancer Patients for Radical Radiation Therapy?
Brief Title: Role of PET CT in Determining Target Volumes in Radiation Therapy for Lung Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Toronto Sunnybrook Regional Cancer Centre (Other)
Collaborators: Ontario Cancer Research Network (Network); Ontario Clinical Oncology Group (OCOG) (Other)
Responsible Party: Yee C. Ung, Sunnybrook Regional Cancer Centre
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 04-may-00142 OCRN; OCRN grant
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2009-02-05 (Estimated); Status verified 2009-02

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-small cell lung cancer; Positron emission tomography; Gross tumor volume; Radiation therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- surgical candidates (Other): surgical candidates who underwent PET CT evaluation
  Interventions: Procedure: Surgical resection

INTERVENTIONS:
Procedure: Surgical resection — pet ct prior to surgery

SUMMARY:
Radiation therapy is an important part of the treatment for lung cancer when treatment intent is for cure. Radiation is a local modality of treatment, that is, it only treats the area that the radiation can target. Therefore it is critical to be able to visualize all the areas of tumor involvement. With current imaging tests such as computed tomography scans (CT), the scans may not be sensitive enough to detect all areas of cancer involvement but with newer imaging tests, such as positron emission tomography (PET), the investigators may be able to better target all the tumor that the CT scan may miss. There are two clinical trials being conducted by the Ontario Clinical Oncology Group (OCOG)looking at PET in lung cancer. This proposal is a companion study to the OCOG PET lung trials. In brief, this study will evaluate the ability of CT alone versus combined PET CT imaging to determine the size of the tumor (or gross tumor volume) along with the tiny extensions of cancer cells (or microscopic extension). The gross tumor volume and its extension as determined by CT or PET CT will then be compared to measurements made on the surgically removed tumor. Treatment with radiation therapy must include all the gross tumor and its extension in order to be successful for cure. If the radiation treatment does not treat all the identified tumor then the chance for cure is lost. There have only been two previous reports of the ability of CT to determine the gross tumor volume and its extension. There are no similar reports using PET CT. This study will be the first of its kind to evaluate how accurate PET CT can be in detecting the gross tumor and its microscopic extension using the surgically removed tumor measurements as the gold standard. If PET CT is able to more accurately determine the tumor volume including its microscopic extension, then this will help oncologists to better treat lung cancer using more accurate radiation treatment volumes.

DETAILED DESCRIPTION:
Radiation therapy is an important component in the curative treatment of non-small cell lung cancer. Targeting of the gross tumor has been facilitated by the use of CT simulation allowing for more accurate delineation of the tumor. In addition multi-modality imaging combining functional and anatomical information have allowed for further refinement in the treatment planning process with significant impact on the planning target volume due to the addition of PET imaging information. PET using 18 F-fluorodeoxyglucose (FDG) allows for more precise detection of tumor since it is a functional image based on glucose metabolism rather than structural abnormalities. Biochemical changes often precede any gross anatomical abnormalities, therefore making PET a very powerful imaging modality. FDG PET has been shown to be more sensitive and specific than CT in the staging of NSCLC.Radical radiation therapy is indicated for early stage NSCLC when the patient is medically inoperable primarily due to co-morbidities. In contrast for locally advanced NSCLC, radical radiation is used as part of induction therapy or in the definitive treatment of NSCLC. In order to avoid a geographical miss with precision radiation therapy, the gross tumor volume (GTV) is outlined and a margin around the GTV is added to incorporate microscopic extension of disease, also known as the clinical target volume (CTV). Standard margins of 1.0 to 1.5 cm are used to encompass the gross tumor, microscopic extent and treatment setup uncertainties.There is surprisingly very little data on what constitutes an adequate margin to encompass the microscopic extent around the gross lung tumor. Studies involving conformal radiation therapy and dose escalation in NSCLC have primarily used an empirical margin to define the CTV. A literature review revealed only two studies evaluating the ability of CT to define the gross tumor and its microscopic extension correlated with histopathological measurements [P Giraud et al 2000, R Chan et al 2001]. The two studies have produced conflicting results with recommended margins being from zero mm to 6-8 mm around the GTV. There have been no studies evaluating the ability of PET to define the size of the gross tumor and its microscopic extension.This is a companion study to the two OCOG PET trials in NSCLC. It will evaluate the ability of CT alone versus PET CT to define the gross tumor and its microscopic extension. The methodology will be based on contouring the GTV with imaging modalities of CT and PET CT and correlating the findings with histopathology.This proposed study will add new information on the ability of combined PET CT to determine the microscopic extension of tumor in NSCLC. While no imaging modality can detect microscopic extension, the newer technology of PET CT may give better resolution over CT alone in the detection of tumor. The strength of this proposal is the required correlation with pathological findings. If PET CT is able to accurately determine the extent of disease, this will have major implications on treatment volumes and subsequent targeting for radiation therapy using 3D conformal radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Surgically resectable non-small cell lung cancer
* Companion clinical trial to OCOG PET Lung trials

Exclusion Criteria:

* Unresectable non-small cell lung cancer
* Unable to undergo PET CT evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2005-10; Primary Completion 2008-06 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Clinical pathological correlation of PET CT with surgically resected NSCLC | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yee C Ung, MD, Principal Investigator — Toronto Sunnybrook Regional Cancer Centre
Locations (1):
- Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario, Canada

REFERENCES:
- [Result] Dahele M, Hwang D, Peressotti C, Sun L, Kusano M, Okhai S, Darling G, Yaffe M, Caldwell C, Mah K, Hornby J, Ehrlich L, Raphael S, Tsao M, Behzadi A, Weigensberg C, Ung YC. Developing a methodology for three-dimensional correlation of PET-CT images and whole-mount histopathology in non-small-cell lung cancer. Curr Oncol. 2008 Oct;15(5):62-9. doi: 10.3747/co.v15i5.349. PMID 19008992